CLINICAL TRIAL: NCT04942106
Title: Biobehavioral Efficacy of the Semi-Elevated Side-Lying Position for Feeding Preterm Infants
Brief Title: Biobehavioral Efficacy of the Semi-Elevated Side-Lying Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston College (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: R21NR019874 (NIH)
Record Dates: First submitted 2021-05-30; First posted 2021-06-28 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Feeding, Bottle; Infant, Premature, Diseases; Behavior, Infant
MeSH Terms: conditions — Bottle Feeding; Infant, Premature, Diseases; Infant Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Side-lying position followed by Supine position (Other): In this arm, infants will be bottle-fed in the side-lying position first followed by the supine position.
  Interventions: Other: Arm 1 - Side-lying position followed by Supine position
- Supine position followed by Side-lying position (Other): In this arm, infants will be bottle-fed in the supine position first followed by the side-lying position.
  Interventions: Other: Arm 2 - Supine position followed by Side-lying position

INTERVENTIONS:
Other: Arm 1 - Side-lying position followed by Supine position — Infants will be observed for two bottle feedings within a 24-hour period when they reach approximately 30-50% oral feeding. In this arm, infants will be bottle-fed in the side-lying position first followed by the supine position. In the side-lying feeding position, the infant will be placed on the caregiver's lap with one ear and hip facing the ceiling at a 45 to 60 degree angle. In the supine feeding position, the infant will be placed facing the caregiver in a reclining position at a 45 to 60 degree angle. In both feeding positions, the infant's head, neck, and upper body will be supported by the caregiver to maintain a neutral straight alignment with the chin tilted down slightly without the neck being extended or in excessive flexion. The infant will also be loosely swaddled with a single blanket so their legs, shoulders, and elbows are supported in a flexed position but with the lower arms free to move.
  Arms: Side-lying position followed by Supine position
Other: Arm 2 - Supine position followed by Side-lying position — Infants will be observed for two bottle feedings within a 24-hour period when they reach approximately 30-50% oral feeding. In this arm, infants will be bottle-fed in the supine position first followed by the side-lying position. In the side-lying feeding position, the infant will be placed on the caregiver's lap with one ear and hip facing the ceiling at a 45 to 60 degree angle. In the supine feeding position, the infant will be placed facing the caregiver in a reclining position at a 45 to 60 degree angle. In both feeding positions, the infant's head, neck, and upper body will be supported by the caregiver to maintain a neutral straight alignment with the chin tilted down slightly without the neck being extended or in excessive flexion. The infant will also be loosely swaddled with a single blanket so their legs, shoulders, and elbows are supported in a flexed position but with the lower arms free to move.
  Arms: Supine position followed by Side-lying position

SUMMARY:
The objective of the proposed research is to conduct a within-subject cross-over trial that will compare the efficacy of the two bottle-feeding positions on physiologic and behavioral responses of preterm infants prior to, during, and after feeding. As an exploratory aim, the investigators will also identify potential infant characteristics associated with the intervention response by evaluating infant sex, maturity level, and/or comorbidity. The two bottle-feeding positions will be the semi-elevated side-lying position (hereafter referred to as side-lying position) and the semi-elevated supine position (hereafter referred to as supine position), which is the traditional feeding position when preterm infants are bottle-fed. The investigators hypothesize that compared to the supine position, the side-lying position will be associated with greater physiologic stability in heart rate, respiratory rate, oxygen saturation, and/or autonomic nervous system regulation during and after feeding. The investigators also hypothesize that compared to the supine position, the side-lying position will be associated with more mature patterns of suck-breathe coordination and/or greater feeding skills.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants who are born at ≤ 35 weeks of GA

Exclusion Criteria:

* Congenital anomaly that may interfere with feeding (e.g., cleft palate or tracheoesophageal fistula)
* Grade IV intraventricular hemorrhage
* Ventilator-dependence beyond 60 days of life
* Inability to orally feed prior to discharge

Max Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Infant physiologic responses to the feeding position - Heart rate (HR) | Up to 30 minutes post-feeding
  HR will be measured for 30 minutes pre-feeding (baseline), feeding, and 30 minutes post-feeding (recovery).
Infant physiologic responses to the feeding position - Respiratory rate (RR) | Up to 30 minutes post-feeding
  RR will be measured for 30 minutes pre-feeding (baseline), feeding, and 30 minutes post-feeding (recovery).
Infant physiologic responses to the feeding position - Oxygen saturation (SaO2) | Up to 30 minutes post-feeding
  SaO2 will be measured for 30 minutes pre-feeding (baseline), feeding, and 30 minutes post-feeding (recovery).
Infant physiologic responses to the feeding position - Heart rate variability (HRV) | Up to 30 minutes post-feeding
  HRV will be measured for 30 minutes pre-feeding (baseline), feeding, and 30 minutes post-feeding (recovery).
Infant physiologic responses to the feeding position - Splanchnic-cerebral oxygen ratio (SCOR) | Up to 30 minutes post-feeding
  SCOR will be measured for 30 minutes pre-feeding (baseline), feeding, and 30 minutes post-feeding (recovery).
Infant behavioral responses to the feeding position - Suck-breathe coordination | 5-30 minutes post-baseline
  Infant behavioral responses will be assessed by the behavioral observation of suck-breathe coordination patterns using Suck-Breath Coordination coding scheme.
Infant behavioral responses to the feeding position - Infant feeding skill | 5-30 minutes post-baseline
  Infant behavioral responses will be assessed by the behavioral observation of infant feeding skill using the Early Feeding Skills (EFS) assessment tool.

SECONDARY OUTCOMES:
Infant characteristics associated with the intervention response - Infant's sex | At enrollment
  Infant's sex (female vs. male)
Infant characteristics associated with the intervention response - Maturity level | At enrollment
  Maturity level will be assessed by gestational age at birth
Infant characteristics associated with the intervention response - Maturity level | At the end of the feeding observation, up to 30 minutes post-feeding
  Maturity level will be assessed by postmenstrual age at the time of study
Infant characteristics associated with the intervention response - Overall severity of illness | At discharge, up to 150 days
  Overall severity illness score will be calculated using the Neonatal Medical Index (range of 1 [least severe] to 5 [most severe])
Infant characteristics associated with the intervention response - Severity of lung disease | At discharge, up to 150 days
  Severity of lung disease will be assessed using diagnostic criteria of bronchopulmonary dysplasia (none, mild, moderate, or severe)

CONTACTS AND LOCATIONS:
Overall Officials: Jinhee Park, PhD, RN, Principal Investigator — Boston College
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
A database will be established to store project data. This data will be free of identifiers that would permit linkages to individual research participants and variables that could lead to deductive disclosure of the identity of individual subjects. Presentations, abstracts, and manuscripts related to the work will also be centrally stored. Once the project is finished and all analyses are complete, it is our intention to make the study dataset available upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The investigators plan to share data starting 6 months after publication upon request.
Access Criteria: Investigators wishing to use the data will submit a written request to the PI and provide a data use agreement with Boston College, stating that the data will be used for scientific purposes. The data and associated documentation will be available to users only under a data-sharing agreement that provides for: 1) a commitment to using the data only for research purposes and not to identify any individual participant; 2) a commitment to securing the data using appropriate computer technology; and 3) a commitment to destroying or returning the data after analyses are completed. There will be no cost for data sharing. Data will be provided to the investigator in an appropriate confidential electronic format.

REFERENCES:
- [Derived] Park J, Thoyre S, Smallcomb J, Mcternan M, Kneeland T. Biobehavioral Efficacy of the Elevated Side-Lying Position for Feeding Preterm Infants: Study Protocol. J Adv Nurs. 2025 May;81(5):2819-2827. doi: 10.1111/jan.16444. Epub 2024 Sep 4. PMID 39231735